CLINICAL TRIAL: NCT04646720
Title: Teleassessment in Neck Pain Patients: an Observational Study
Brief Title: Teleassessment in Neck Pain
Acronym: Teleneck
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Other Study IDs: DF0092UG
Record Dates: First submitted 2020-11-13; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Neck Pain; Assessment, Self; Kinesiophobia
MeSH Terms: conditions — Neck Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neck pain patients: Patients with neck pain evaluated with new technologies and face-to-face

SUMMARY:
New technologies have improved the aproach of patients with different pathologies. Neck pain is a prevalent pathology in physical therapy clinics. Evaluating patients with an electronical device could decrease the services saturation and the proffesionals overload.

ELIGIBILITY:
Inclusion Criteria:

* Presence of neck pain
* Between 18 and 65 years
* Accepted to sign the informed consent

Exclusion Criteria:

* Cognitive impairment.
* Traumatic accidents.
* Other orthopedic or neurologic pathology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic neck pain
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in range of movement | Baseline
  Changes in range of movement were measured with goniometry and expressed in degrees.
Changes in trigger points | Baseline
  Changes in trigger points were measured following the Travels and Simons protocol in the trapezius, suboccipitalis, scalenes and sternocleidomastoid muscles. The number od trigger points found was registered.
Changes in neck endurance (anterior) | Baseline
  Changes in neck endurance were measured using an endurance test for the anterior neck muscles. The time performing the test was registered.
Changes in neck endurance (posterior) | Baseline
  Changes in neck endurance were measured using an endurance test for the posterior neck muscles. The time performing the test was registered.
Changes in quality of life | Baseline
  Changes in quality of life were measured using the Euroqol 5dimensions which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. It also includes a visual analogue scale to report the health status from 0 to 100.
Changes in quality of life (Visual Analogue Scale) | Baseline
  Changes in quality of life were measured using the Euroqol 5dimensions which comprises a visual analogue scale to report the health status from 0 to 100.

SECONDARY OUTCOMES:
Changes in kinesiophobia | Baseline
  Changes in kinesiophobia were measured using the Tampa Scale for Kinesiophobia (TSK) which is one of the most frequently employed measures for assessing pain-related fear in pain patients.
Changes in functionality | Baseline
  Changes in functionality were measured using the World Health Organization Disability Assessment Schedule, WHODAS-2, which provides a global measure of disability and 7 domain-specific scores.

IPD SHARING:
Plan to Share IPD: No